CLINICAL TRIAL: NCT02238652
Title: Improving Quality of Life in Nursing Home Residents: A Cluster Randomized Clinical Trial of Efficacy (The KOSMOS Study)
Brief Title: Improving Quality of Life in Nursing Home Residents: A Cluster Randomized Clinical Trial of Efficacy
Acronym: KOSMOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: The Research Council of Norway (Other); Rebekka Ege Hegemanns legat (Unknown); Helse Stavanger HF (Other Government); University of Oslo (Other); King's College London (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Bettina Husebo, MD, assoc prof., University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 222113
Record Dates: First submitted 2014-07-07; First posted 2014-09-12 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2014-09

CONDITIONS: Quality of Life
Keywords: Nursing homes; Dementia; Quality of Life; Geriatrics; Aged; Activities of Daily Living; Pain; Pain management; Advance Care Planning; Patient Safety; Costs and Cost Analysis; Medication Errors; Medical Order Entry Systems; Medication Reconciliation; Medication Therapy Management; Depression; Psychotropic Drugs; Informed Consent; Presumed Consent; Anxiety; Apathy; Hospitalization; Mortality
MeSH Terms: conditions — Dementia; Pain; Agnosia; Depression; Anxiety Disorders; Lethargy | interventions — Advance Care Planning; Therapeutics; Medication Review; Occupational Therapy; Safety; Patient Safety

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Intervention (Active Comparator): Communication Systematic Pain Assessment and Treatment Medication Review Occupational therapy Safety
  Interventions: Behavioral: Communication; Behavioral: Systematic Pain Assessment and Treatment; Behavioral: Medication Review; Behavioral: Occupational therapy; Behavioral: Safety

INTERVENTIONS:
Behavioral: Communication — A preparation process before the patient become incapable of participating in life prolonging decisions
  Other Names: advance care planning
  Arms: Intervention
Behavioral: Systematic Pain Assessment and Treatment — Assess pain with MOBID-2 Pain Scale and thereby improve pain management in dementia.
  Other Names: MOBID-2
  Arms: Intervention
Behavioral: Medication Review — An individual and systematic review of medication prescriptions to identify possible harmful drug effects and to reduce the use of psychotropic drugs.
  Arms: Intervention
Behavioral: Occupational therapy — Increase individual activities, based on function, personal interest and personality by educating the staff on these elements.
  Arms: Intervention
Behavioral: Safety — Focusing on developing a culture where staff has an active and constant awareness of how to prevent adverse events and a commitment to safety.
  Other Names: patient safety
  Arms: Intervention

SUMMARY:
Improving quality of life (QoL) in residents of nursing homes:

A cluster randomized clinical trial of efficacy - The KOSMOS study.

COSMOS (COmmunication (Advance Care Planning - ACP), Systematic pain assessment and treatment, Medication review, Occupational therapy, and Safety) is a practical intervention aimed to improve clinical and psychiatric challenges in NH patients. The COSMOS intervention combines the most effective research results to improve staff competence and patients' mental health, safety, QoL. We also aim to reduce psychotropic drug use and costs.

DETAILED DESCRIPTION:
Background: Nursing home (NH) patients have complex mental health problems, disabilities and social needs, compounded by widespread prescription of psychotropic drugs. To preserve their dignity and quality of life is an important goal of our society. This can only be achieved within NHs that offer high competent conditions of treatment and care.

Research questions and hypotheses:

1. Will the implementation of a communication and end-of-life decision making process have impact on interactions between patients, staff and family? We hypothesize that ACP will improve the interactions between patients, staff and family, and satisfaction in relatives and thereby improve the quality of life NH patients.
2. Is the KOSMOS capable to affect agitation and aggression and reduce medication e.g. psychotropics in NH patient? We hypothesize that KOSMOS will significantly reduce agitation and aggression, the total amount of medication, and psychotropic drug use.
3. What combination of interventions will give the broadest benefit, and could be delivered as a routine intervention as part of NH practice? We hypothesize that the comprehensive KOSMOS approach improves QoL and makes positive changes in NH practice.
4. What other types of advantages are expected? We hypothesize that KOSMOS is a cost-effective approach, with potential to increase the safety and reduce mortality in NH patients.

Method: The KOSMOS intervention combines the most effective research results to improve staff competence, and patients' mental health, safety, QoL, and to reduce psychotropic drug use and costs. The efficacy testing of KOSMOS includes systematic literature review, a pilot study, a 9-month randomized control trial (RCT), and a dissemination plan. Data collection will take place at baseline, months 4, and 9. The intervention entails provision of staff training, study guidelines and manuals. NHs will be randomized to either KOSMOS or current best practice. We will include 38 NH long-term-care (LTC) wards (normally just one ward per NH) in Bergen, Stavanger, Oslo/Bærum, Sarpsborg and Sogn and Fjordane. In total 310 patients ≥65 years will be recruited from these wards

Primary and secondary outcome measures: Quality of life in late stage dementia (QUALID), QUALIDEM, EQ-5-D; Neuropsychiatric Inventory - NH edition (NPI-NH); Activities of Daily Living (ADL); Cornell; Mobilization - Observation - Behaviour - Intensity - Dementia 2 (MOBID-2); drug use; drug-related problems, START; STOP; cost-utility analysis (RUD-FOCA); hospital admission; and mortality, ActiWatch; Log registration of NH activities; Relatives satisfaction with conducted KOSMOS elements

Statistical analyses: include characteristics between 2 groups (Chi square, Mann-Whitney U), ANCOVA, ICC and p-values for each time-point and outcomes.

National and international collaboration: National collaboration between researchers at the Universities of Bergen, Oslo, and Stavanger is established. Internationally, colleagues from the EU COST-Action TD1005, Karolinska University, Stockholm and Kings College, London are engaged in this RCT.

Funding: The employment of two PhD-candidates (100%) and one post-doctoral fellow (50%) received funding by the Norwegian Research Council (Sponsor's Protocol Code: 222113) in 2012.

ELIGIBILITY:
Inclusion Criteria:

* Resident in long time care ward in Bergen, Bærum, Sarpsborg, Kvam, Fjell, Sund, Askøy and Øygarden

Exclusion Criteria:

* Dying patients with reduced consciousness at baseline
* Active Schizophrenia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 560 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric symptoms | 9 months
  Depression, anxiety an apathy will be assessed by the Neuropsychiatric Inventory - Nursing Home version (NPI-NH).
Quality of life | 9 months
  Assessing quality of life by Qualidem, QUALID and EQ-5D.

SECONDARY OUTCOMES:
Activities of daily living | 9 months
  Assessed by ADL index (range 0-18).
Mood or depression | 9 months
  Assessed by Cornell Depression Scale (range 0-38)
Pain | 9 months
  Assessed by Mobilisation-Observation-Behaviour-Intensity-Dementia (MOBID-2) Pain Scale (range 0-10)
Medication review | 9 months
  Use of medication in number of people and dose, especially use of psychotropic drugs
Drug-related problems | 9 months
  number of drug-drug-interactions using interactions database, number of drugs prescribed, number of anticholinergics prescribed, number of patients prescribed pain-medication with no pain on the MOBID-2 pain scale, number of patients with anti depressants with a low cornell depression rating scale in dementia.
Admission to hospital and mortality | 9 months
  Questionnaire asking nurses wether the patient has been admitted to the hospital at month 4 and month 9.
Cost-effectiveness | 9 months
  Resource use will be registered by Resource use in dementia - formal care (RUD-FOCA)
Cost of medication | 9 months
  Cost-utility analysis will be performed
Measure of activity | 9 months
  ActiWatch to register sleep and activity
Nursing home activity | 9 months
  Log registration of NH activities
Relatives satisfaction with conducted KOSMOS elements | 9 months
  Relatives satisfaction with conducted KOSMOS elements with questionary

OTHER OUTCOMES:
Implementation indicators | 9 months
  Assessment of the quality of the implementation on each intervention by monthly visits and phone calls and review of the manuals.

CONTACTS AND LOCATIONS:
Overall Officials: Bettina S. Husebø, MD, PhD, Study Director — University of Bergen; Elisabeth Flo, PysD, PhD, Principal Investigator — University of Bergen; Irene Aasmul, Master, Principal Investigator — University of Bergen; Christine Gulla, MD, Principal Investigator — University of Bergen; Torstein Habiger, Principal Investigator — University of Bergen; Tony Elvegaard, Principal Investigator — University of Bergen
Locations (32):
- Norway (32):
  - Solvik, Baerum, Akershus
  - Donski Bo og behandlingssenter, Baerum, Akershus
  - Mariehaven Bo og behandlingssenter, Baerum, Akershus
  - Berger Bo og Behandlingssenter, Baerum, Akershus
  - Kolaashjemmet Bo og Behandlingssenter, Baerum, Akershus
  - Gullhaug Bo og behandlingssenter, Baerum, Akershus
  - Osteraas Bo og behandlingssenter, Baerum, Akershus
  - Solbakken Bo og Behandlingssenter, Baerum, Akershus
  - Lønnås Bo og Rehabsenter, Baerum, Akershus
  - Nordraaksvei bo og behandlingssenter, Baerum, Akershus
  - Stabaekktunet Bo og behandlingssenter, Baerum, Akershus
  - Stabekk Bo og Behandlingssenter, Baerum, Akershus
  - Ask bo og omsorgssenter, Askøy
  - Arna helseheim, Bergen
  - Frieda Fasmers minne, Bergen
  - Gullstøltunet Sykehjem, Bergen
  - Hospitalet Betanien, Bergen
  - Lyngbøtunet Bo og servicesenter, Bergen
  - Slettebakken menighets eldresenter, Bergen
  - University of Bergen, Bergen
  - Strandebarmheimen, Kvam
  - Toloheimen, Kvam
  - Øysteseheimen, Kvam
  - Borgen sykehjem, Sarpsborg
  - Eplehagen bofellesskap, Sarpsborg
  - Haugvoll sykehjem, Sarpsborg
  - Helsehuset, Sarpsborg
  - Kurland, Sarpsborg
  - Tingvoll sykehjem, Sarpsborg
  - Valaskjold omsorgssenter, Sarpsborg
  - Sundheimen, Sund
  - Tednebakkane omsorgssenter, Øygarden

REFERENCES:
- [Background] Husebo BS, Flo E, Aarsland D, Selbaek G, Testad I, Gulla C, Aasmul I, Ballard C. COSMOS--improving the quality of life in nursing home patients: protocol for an effectiveness-implementation cluster randomized clinical hybrid trial. Implement Sci. 2015 Sep 15;10:131. doi: 10.1186/s13012-015-0310-5. PMID 26374231
- [Derived] Vislapuu M, Berge LI, Angeles RC, Kjerstad E, Mannseth J, Achterberg WP, Husebo BS. Factors associated with formal and informal resource utilization in nursing home patients with and without dementia: cross-sectional analyses from the COSMOS trial. BMC Health Serv Res. 2022 Nov 2;22(1):1306. doi: 10.1186/s12913-022-08675-y. PMID 36324159
- [Derived] Flo-Groeneboom E, Elvegaard T, Gulla C, Husebo BS. The longitudinal association between the use of antihypertensive medications and 24-hour sleep in nursing homes: results from the randomized controlled COSMOS trial. BMC Geriatr. 2021 Jul 18;21(1):430. doi: 10.1186/s12877-021-02317-4. PMID 34275457
- [Derived] Gedde MH, Husebo BS, Mannseth J, Kjome RLS, Naik M, Berge LI. Less Is More: The Impact of Deprescribing Psychotropic Drugs on Behavioral and Psychological Symptoms and Daily Functioning in Nursing Home Patients. Results From the Cluster-Randomized Controlled COSMOS Trial. Am J Geriatr Psychiatry. 2021 Mar;29(3):304-315. doi: 10.1016/j.jagp.2020.07.004. Epub 2020 Jul 11. PMID 32753339
- [Derived] de Jong-Schmit BEM, Poortvliet RKE, Bohringer S, Bogaerts JMK, Achterberg WP, Husebo BS. Blood pressure, antihypertensive medication and neuropsychiatric symptoms in older people with dementia: The COSMOS study. Int J Geriatr Psychiatry. 2021 Jan;36(1):46-53. doi: 10.1002/gps.5388. Epub 2020 Oct 8. PMID 32748494
- [Derived] Gulla C, Flo E, Kjome RLS, Husebo BS. Implementing a novel strategy for interprofessional medication review using collegial mentoring and systematic clinical evaluation in nursing homes (COSMOS). BMC Geriatr. 2019 May 7;19(1):130. doi: 10.1186/s12877-019-1139-6. PMID 31064365
- [Derived] Habiger TF, Achterberg WP, Flo E, Husebo BS. Psychosis symptoms in nursing home residents with and without dementia-Cross-sectional analyses from the COSMOS study. Int J Geriatr Psychiatry. 2019 May;34(5):683-691. doi: 10.1002/gps.5067. Epub 2019 Mar 4. PMID 30706561
- [Derived] Aasmul I, Husebo BS, Sampson EL, Flo E. Advance Care Planning in Nursing Homes - Improving the Communication Among Patient, Family, and Staff: Results From a Cluster Randomized Controlled Trial (COSMOS). Front Psychol. 2018 Dec 4;9:2284. doi: 10.3389/fpsyg.2018.02284. eCollection 2018. PMID 30564163
- [Derived] Aasmul I, Husebo BS, Flo E. Description of an advance care planning intervention in nursing homes: outcomes of the process evaluation. BMC Geriatr. 2018 Jan 25;18(1):26. doi: 10.1186/s12877-018-0713-7. PMID 29370766
- [Derived] Blytt KM, Bjorvatn B, Husebo B, Flo E. Clinically significant discrepancies between sleep problems assessed by standard clinical tools and actigraphy. BMC Geriatr. 2017 Oct 27;17(1):253. doi: 10.1186/s12877-017-0653-7. PMID 29078755
- See also: Centre for Elderly and Nursing Home Medicine — http://www.uib.no/sefas